CLINICAL TRIAL: NCT03916263
Title: Compare Weight Loss and Metabolic Improvements Using a Low Starch Dietary Education Program vs. Traditional Treatment for Polycystic Ovary Syndrome (PCOS)
Brief Title: Low Starch Dietary Education Program vs. Traditional Treatment for PCOS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L18-147
Record Dates: First submitted 2019-01-21; First posted 2019-04-16 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: PCOS; Diet Modification; Metabolism; Nutrition Disorders
Keywords: PCOS; Diet; Video Instruction
MeSH Terms: conditions — Nutrition Disorders | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Prospective Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Traditional Treatment (Experimental): Participant receives recommendations for caloric intake, exercise and prescription for metformin if indicated
  Interventions: Drug: Metformin
- One-On-One Low Starch Dietary Instruction (Other): Participant receives One-On-One Low Starch Dietary Instruction from Study Collaborator
  Interventions: Other: One-On-One Dietary Instruction
- Low Starch Dietary Instruction by Video (Other): Participant receives Low Starch Dietary Instruction by Video Link
  Interventions: Other: Video Dietary Instruction

INTERVENTIONS:
Drug: Metformin — Traditional care including diet, exercise and metformin
  Other Names: Traditional care
  Arms: Traditional Treatment
Other: One-On-One Dietary Instruction — Participant receives one-on-one dietary counseling from study personnel
  Arms: One-On-One Low Starch Dietary Instruction
Other: Video Dietary Instruction — Participant receives video dietary instruction
  Arms: Low Starch Dietary Instruction by Video

SUMMARY:
Compare weight loss and metabolic parameters in patients using a low starch dietary education program vs. traditional treatment (i.e., prescribing metformin, low calorie diet and exercise) for health improvement in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common gynecologic condition diagnosed by the presence of irregular menstruation, high androgen levels and polycystic appearing ovaries by ultrasound. PCOS affects approximately 5 million women of reproductive age in the United States and is associated with increased risk of obesity, diabetes, cardiovascular disease, cancer and infertility. Women with PCOS are at 5- to 10-fold risk of developing type 2 diabetes and are diagnosed on average 30 years sooner than women without PCOS. Historically, high insulin levels worsen symptoms of PCOS and make weight loss very difficult despite the patient's best efforts. Research shows that carbohydrates from dairy and starch-based foods have greater insulin-producing properties than carbohydrates from non-starchy vegetables and fruits. The purpose of this study is to compare metabolic parameters in patients using a low starch dietary education program vs. traditional treatment (i.e., prescribing metformin, low calorie diet and exercise) for health improvement in women with PCOS.

In the investigator's previous work, study participants received approximately 1.5 hours of one-on-one dietary instruction by a Registered Dietitian. Dietary instruction included review of a list of foods that participants could eat with no restrictions as well as a list of foods to avoid, i.e. grains and dairy products. Study participants, all of whom were overweight or obese, achieved an average weight loss of 18.9 pounds in 8 weeks. In addition, study participants demonstrated improvements in triglycerides, total and free testosterone and in clinical hair growth scores. This study will investigate whether the same positive results might be achieved using a web-based written and video program for dietary guidance. If successful, the dietary video instructions may potentially benefit a large number of women by providing health care providers with a practical and affordable method to provide dietary instructions to their patients with PCOS, especially in areas where access to a Registered Dietitian is limited.

The goal of this prospective, randomized, controlled, clinical trial is to develop a practical, clinically useful web-based tool for health care providers to educate their patients on an optimal eating plan to manage PCOS.

AIM:

1.Compare weight loss and metabolic parameters in patients using a low starch dietary education program vs. traditional treatment (i.e., prescribing metformin, low calorie diet and exercise) for health improvement in women with PCOS.

METHODS:

Sixty overweight women with PCOS will be recruited to participate in an 8-week low starch diet with pre- and post-study measurements of weight, body mass index, waist to hip ratio, fasting glucose and insulin, complete lipid panel, free and total testosterone, and hemoglobin A1c. Patients will be randomized 1:1 to receive web-based instruction for a low starch diet or to receive face to face nutritional and diet information, or to receive a traditional care plan (metformin if indicated, low calorie diet, and exercise).

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-45
* BMI of >25 but < 45
* PCOS
* Access to a computer/phone/electronic device with internet connection.

Exclusion Criteria:

* Pregnancy
* Abnormal thyroid stimulating hormone (TSH)
* Hyperprolactinemia
* adrenal hyperplasia
* Cushing's disease Ovarian and adrenal tumors. Previous diagnosis of diabetes. History of eating disorder History of surgical weight loss procedure Persons with an inability to give informed consent Persons unable/unwilling to exercise or to prepare their own food

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Weight | 8 weeks
  Weight
BMI | 8 weeks
  BMI

SECONDARY OUTCOMES:
waist to hip ratio | 8 weeks
  waist to hip ratio
fasting glucose | 8 weeks
  fasting glucose
fasting insulin | 8 weeks
  fasting insulin
cholesterol | 8 weeks
  cholesterol
testosterone | 8 weeks
  testosterone
hemoglobin A1c | 8 weeks
  hemoglobin A1c

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Phy, DO, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech Health Science Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Will post to Clinical Trials
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: 2 years